CLINICAL TRIAL: NCT01368653
Title: Evaluation of Learning-Theory-Based Smoking Cessation Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Danielle E. McCarthy, Ph.D., Associate Professor, Rutgers University
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA026511; 1R21DA026511-01A1 (NIH)
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Results first posted 2014-11-18 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-03

CONDITIONS: Nicotine Dependence
Keywords: Tobacco; Smoking; Smoking Cessation; Tobacco Dependence; Tobacco Use; Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Smoking Cessation; Tobacco Use | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard treatment (Active Comparator): In this arm, smokers receive a 6-week supply of 21-mg nicotine patches and 4 15-minute individual smoking cessation counseling sessions to help them quit smoking
  Interventions: Behavioral: Standard treatment
- Standard treatment+practice quitting (Experimental): In this arm, participants receive standard treatment (a 6-week supply of 21-mg nicotine patches and 4 15-minute individual smoking cessation counseling session) and an experimental treatment that involves practice quitting 7 times prior to a target quit date (for 4-12 hours per day) and returning to smoking by puffing smoke without inhaling.
  Interventions: Behavioral: Standard treatment+practice quitting
- Very low nicotine cigarettes (Experimental): In this condition, smokers from both the Standard treatment and the Standard treatment+practice quitting arms who have smoked in the last 7-days at a 4-week post-target-smoking-cessation-date follow-up interview may be randomly assigned to this group. Those assigned to this group will receive a 6-week supply of cigarettes that contain tobacco with very low levels of nicotine (in regular or menthol flavors) to smoke instead of regular cigarettes containing nicotine. This treatment is designed to help people stop smoking after slipping (returning to smoking) during an attempt to stop smoking
  Interventions: Drug: Very low nicotine cigarettes
- Advice and encouragement only (No Intervention): In this condition, smokers from both the Standard treatment and the Standard treatment+practice quitting arms who have smoked in the last 7-days at a 4-week post-target-smoking-cessation-date follow-up interview may be randomly assigned to this condition. Those in this arm will receive advice and encouragement to try to stop smoking again after they have slipped (returned to smoking) during a stop smoking attempt.

INTERVENTIONS:
Behavioral: Standard treatment — Standard treatment includes a 6-week supply of 21-mg nicotine patches and 4 15-minute individual smoking cessation counseling sessions to help smokers quit smoking
  Other Names: Nicotine patch
  Arms: Standard treatment
Behavioral: Standard treatment+practice quitting — This intervention includes standard treatment (a 6-week supply of 21-mg nicotine patches and 4 15-minute individual smoking cessation counseling session) and an experimental treatment that involves practice quitting 7 times prior to a target quit date (for 4-12 hours per day) and returning to smoking by puffing smoke without inhaling
  Other Names: Nicotine patch
  Arms: Standard treatment+practice quitting
Drug: Very low nicotine cigarettes — This intervention will be offered to a subset of smokers from both of the other study arms. To be eligible for this intervention, participants must be smoking at the follow-up interview conducted four weeks after a target quit day in the two arms listed above. Tobacco cigarettes containing very low levels of nicotine (.016-.019 mg in smoke from the cigarettes). These are to be smoked no more often than a smoker normally smokes regular cigarettes and for no longer than 6 weeks.
  Arms: Very low nicotine cigarettes

SUMMARY:
This clinical trial tested whether a new treatment designed to help smokers prepare to quit smoking by practicing quitting several times helped more smokers quit and stay quit than standard treatment with nicotine patch and smoking cessation counseling. The practice quitting treatment tested involved quitting for progressively longer periods of time tailored to individual patterns of smoking. This clinical trial also tested whether non-nicotine cigarettes can help smokers become smoke free after slipping during a stop smoking attempt.

DETAILED DESCRIPTION:
* Participants in this study are randomized to one of two treatments conditions prior to a target quit date.

  * One-half of participants will be randomly assigned to receive standard smoking cessation treatment comprising a 6-week supply of 21-mg nicotine patches and 4 individual smoking cessation counseling sessions.
  * The other one-half of participants will be randomly assigned to receive standard treatment (patch and counseling, as above) plus to practice quitting 7 times over the 2.5 weeks leading up to a quit attempt. Practice quitting will involve not smoking for a period of time tailored to each individual's smoking pattern.
* All participants are asked to attend a 2-hour orientation session, complete 8 brief (5-minute) telephone calls and 9 longer(20-minute) telephone surveys over 3.5 weeks, attend a 30-minute office visit, and complete two 15-minute follow-up calls.
* All participants are also asked to report on their emotions, thoughts, and behaviors 3 times per day for 24 days using cellular telephones.
* Participants receive compensation for office visits, study telephone calls, cellular telephone reports, and follow-up interviews.
* All participants will receive nicotine patches and one-on-one counseling (delivered over the phone and in person).
* Some participants will be eligible for a second phase of treatment after a 4-week follow-up interview.

  * One-half of people eligible for this phase of the study will be randomly assigned to receive a supply of non-nicotine cigarettes to smoke for up to 6 weeks. The non-nicotine cigarettes are designed to help break the habit of smoking and to help smokers return to being smoke-free after smoking regular cigarettes.
  * The other one-half of eligible smokers will be randomly assigned to not receive these non-nicotine cigarettes.
  * All smokers eligible for this phase of the study will be asked to complete cellular telephone reports about their mood, thoughts, and behaviors for 14 days beginning 4.5 weeks after a target stop-smoking date. Compensation will be provided for completing these cellular telephone phone reports.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Smoke cigarettes daily
* Motivated to quit smoking
* Able to read and write English
* Willing and able to complete study visits and cell phone calls

Exclusion Criteria:

* Pregnancy, breastfeeding, planning on becoming pregnant during the study
* Recent heart attack or heart surgery, heart disease, unstable angina
* Allergy to adhesives
* Past negative reactions to nicotine patch
* Serious skin conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle E McCarthy, Ph.D., Principal Investigator — Rutgers University
Locations (1):
- Rutgers University Institute for Health, Health Care Policy, and Aging Research, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between June 12, 2012 and May 24, 2013 through community-wide recruitment including direct mail, flyers, and radio advertising.
Pre-assignment Details: Randomization was in 2 phases; 1: participants who met inclusion/exclusion criteria were randomized to either standard treatment or standard treatment plus practice quitting; in phase 2, smokers who smoked between weeks 3 and 4 post-quit were randomly assigned to either receive advice only, or advice plus very low nicotine cigarettes.
Period: Overall Study
Arm/Group | Standard Treatment | Standard Treatment+Practice Quitting
Started | 47 | 46
Completed 4-week Follow-up | 44 | 37
Smoked in Past 7 Days at 4-weeks | 29 (The first 40 who smoked between weeks 3 and 4 post-quit were eligible for Phase 2 (VLNC vs. Advice)) | 20 (The first 40 who smoked between weeks 3 and 4 post-quit were eligible for Phase 2 (VLNC vs. Advice))
Randomized to Phase 2 | 21 (The first 40 who smoked between weeks 3 and 4 post-quit were eligible for Phase 2 (VLNC vs. Advice)) | 19 (The first 40 who smoked between weeks 3 and 4 post-quit were eligible for Phase 2 (VLNC vs. Advice))
Randomized to VLNC in Phase 2 | 11 (VLNC=6-week supply of Very Low Nicotine Cigarettes plus Advice to Quit (vs. Advice Only)) | 9 (VLNC=6-week supply of Very Low Nicotine Cigarettes plus Advice to Quit (vs. Advice Only))
Randomized to Advice Only in Phase 2 | 10 | 10
Completed | 41 | 37
Not Completed | 6 | 9

BASELINE CHARACTERISTICS:
Population: The total number of participants in the sample was 93. The 40 participants randomly assigned to Very low nicotine cigarettes or Advice and encouragement only were a subset of the 93 participants randomly assigned to initial experimental conditions (Standard treatment or Standard treatment+practice quitting) if still smoking at 4-week follow-up.
Groups:
- Standard Treatment: In this arm, smokers received a 6-week supply of 21-mg nicotine patches and 4 15-minute individual smoking cessation counseling sessions to help them quit smoking
  Standard treatment: Standard treatment included a 6-week supply of 21-mg nicotine patches and 4 15-minute individual smoking cessation counseling sessions to help smokers quit smoking
- Standard Treatment+Practice Quitting: In this arm, participants received standard treatment (a 6-week supply of 21-mg nicotine patches and 4 15-minute individual smoking cessation counseling session) and an experimental treatment that involves practice quitting 7 times prior to a target quit date (for 4-12 hours per day) and returning to smoking by puffing smoke without inhaling.
  Standard treatment+practice quitting: This intervention included standard treatment (a 6-week supply of 21-mg nicotine patches and 4 15-minute individual smoking cessation counseling session) and an experimental treatment that involves practice quitting 7 times prior to a target quit date (for 4-12 hours per day) and returning to smoking by puffing smoke without inhaling
- Total: Total of all reporting groups
Arm/Group | Standard Treatment | Standard Treatment+Practice Quitting | Total
Number analyzed (Participants) | 47 | 46 | 93
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 45 | 90
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.13 (14.27) | 48.41 (10.36) | 47.76 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 23 | 22 | 45
Region of Enrollment [Number; unit: participants]
  United States | 47 | 46 | 93

OUTCOME MEASURES:

1. Primary Outcome: 4-week Abstinence
Description: 7-day point prevalence abstinence captures whether participants have used tobacco in the past 7 days at the 4-week post-quit follow-up (i.e., whether any tobacco use occurred in the 4th week of the quit attempt).
Time Frame: 4 weeks
Measure: Number; unit: participants
Groups:
- Standard Treatment+Practice Quitting: In this arm, participants received standard treatment (a 6-week supply of 21-mg nicotine patches and 4 15-minute individual smoking cessation counseling session) and an experimental treatment that involved practice quitting 7 times prior to a target quit date (for 4-12 hours per day) and returning to smoking by puffing smoke without inhaling.
  Standard treatment+practice quitting: This intervention included standard treatment (a 6-week supply of 21-mg nicotine patches and 4 15-minute individual smoking cessation counseling session) and an experimental treatment that involved practice quitting 7 times prior to a target quit date (for 4-12 hours per day) and returning to smoking by puffing smoke without inhaling
Arm/Group | Standard Treatment | Standard Treatment+Practice Quitting
Number analyzed (Participants) | 47 | 46
participants
  Abstinent (no smoking reported in past 7 days) | 15 | 17
  Smoking (any cigarettes in past 7 days) | 29 | 20
  Lost to 4-week follow-up | 3 | 9

2. Secondary Outcome: 10-week Abstinence
Description: This captures whether any tobacco use occurred in the past 7 days at the 10-week follow up (i.e., whether any tobacco use occurred in the 10th week of the quit attempt), as reported by participants in a timeline follow-back telephone interview and confirmed by a follow-up expired carbon monoxide reading less than or equal to 8 parts per million.
Time Frame: 10 weeks
Measure: Number; unit: participants
Groups:
- Very Low Nicotine Cigarettes: Smokers who had smoked in the last 7 days at the 4-week telephone follow-up interview (N=40) were randomly assigned to either this condition (n=20) or a smoking cessation advice and encouragement control condition (n=20) at the 4-week follow-up. In this condition, smokers received a 6-week supply of cigarettes that contained tobacco with very low levels of nicotine (in regular or menthol flavors) to smoke instead of regular cigarettes containing nicotine. This treatment was designed to help people stop smoking after slipping (returning to smoking) during an attempt to stop smoking
  Very low nicotine cigarettes: Tobacco cigarettes containing very low levels of nicotine (.016-.019 mg in smoke from the cigarettes). These were to be smoked no more often than a smoker normally smokes regular cigarettes and for no longer than 6 weeks.
- Advice and Encouragement Only: Smokers who had smoked in the last 7 days at the 4-week telephone follow-up interview (N=40) were randomly assigned to either this condition (n=20) or a very-low-nicotine-cigarette condition (n=20) at the 4-week follow-up. In this control condition, smokers received advice and encouragement to try to stop smoking again at the 4-week follow-up after they slipped (returned to smoking) during a stop smoking attempt.
Arm/Group | Standard Treatment | Standard Treatment+Practice Quitting | Very Low Nicotine Cigarettes | Advice and Encouragement Only
Number analyzed (Participants) | 47 | 46 | 20 | 20
participants
  Abstinent (no smoking past 7 days) CO-confirmed | 5 | 11 | 2 | 1
  Smoking (any cigarettes in past 7 days) | 36 | 26 | 17 | 19
  Lost to 10-week follow-up | 6 | 9 | 1 | 0

3. Secondary Outcome: Mediators of Treatment Effects: Confidence in Quitting in the Weeks Leading up to the Target Quit Date
Description: Emotional, mental, and behavioral measures that may help explain treatment effects on tobacco use outcomes will be assessed intensively in the three weeks leading up to a quit attempt and the first week of a quit attempt to examine mediators (confidence in quitting) of the first phase treatment. These repeated measures will be analyzed to see if treatment affects them and if they predict smoking behavior. Confidence related to quitting to for good was rated on a 5-point scale where 1=definitely not confident and 5=definitely confident.
Time Frame: 3 weeks pre-quit
Population: Participants who quit for at least 1 day in the first 2 weeks after the target quit date.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Standard Treatment | Standard Treatment+Practice Quitting
Number analyzed (Participants) | 37 | 37
units on a scale | 4.39 (0.14) | 3.70 (0.22)

4. Secondary Outcome: Prolonged Abstinence
Description: This outcome measures whether regular smoking (7 days in a row) occurred between the 4th and 10th weeks of the quit attempt.
Time Frame: 10 weeks
Measure: Number; unit: participants
Arm/Group | Standard Treatment | Standard Treatment+Practice Quitting | Very Low Nicotine Cigarettes | Advice and Encouragement Only
Number analyzed (Participants) | 47 | 46 | 20 | 20
participants
  Abstinent (no smoking 7 days in a row) | 14 | 20 | 1 | 6
  Smoking (7 days in a row) | 27 | 17 | 18 | 14
  Lost to 10-week follow-up | 6 | 9 | 1 | 0

ADVERSE EVENTS:
Time Frame: All participants were asked to report any changes in their health at every live assessment contact with them following the initiation of treatment (a total of 19 contacts over the course of 12 weeks).
Description: Assessment was systematic in that all researchers were trained to provide a standardized prompt "Have you noticed any changes in your health since we last spoke with you?" at every live assessment call or visit during the study.
Arm/Group | Standard Treatment | Standard Treatment+Practice Quitting | Very Low Nicotine Cigarettes | Advice and Encouragement Only
Serious Adverse Events (participants affected / at risk) | 3/47 | 4/46 | 2/20 | 1/20
Other Adverse Events (participants affected / at risk) | 29/47 | 22/46 | 10/20 | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment (N=47) | Standard Treatment+Practice Quitting (N=46) | Very Low Nicotine Cigarettes (N=20) | Advice and Encouragement Only (N=20)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Tooth abscess requiring emergency surgery and overnight hospitalization
Upper GI tract disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Participant reported that he was hospitalized for severe upper gastrointestinal tract problems, had an endoscopy, and was prescribed new medication. Participant was not on study medication at the time of his symptoms or hospitalization.
Broken toe (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant reported an injury that broke a toe and said that she was hospitalized overnight for observation. Participant reported using study medication (nicotine patch) at the time of the injury.
Chest pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Participant reported experiencing chest pain; she went to an emergency dept., had an ECG, and cardiac catheterization before leaving with a negative diagnosis for cardiac disorder. She was given esomeprazole and sucralfate and an endoscopy order.
Leg and back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Participant reported leg and back pain worsening over three months that prompted an emergency dept. visit and hospitalization for MRI and plethysmography; left with pain medication.
Bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant experienced nausea, vomiting, abdominal pain; was admitted to hospital, diagnosed with a bowel obstruction, treated, and released after 5 days.
Respiratory distress, diabetes, and dehydration (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — At follow-up, participant reported 4 emergency dept. visits and hospitalization for varied symptoms (cough, chills, nausea, abdominal pain, headache) and said she was treated for dehydration, had her insulin for DM-II adjusted, and had a procedure.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment (N=47) | Standard Treatment+Practice Quitting (N=46) | Very Low Nicotine Cigarettes (N=20) | Advice and Encouragement Only (N=20)
Respiratory infection, congestion, or illness (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 7 (7) | 3 (3) | 4 (4) — Symptoms of nasal or sinus congestion, sore throat, asthma (in previously diagnosed individuals), and mild shortness of breath.
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 7 (7) | 4 (4) | 4 (4) — Cough, whether dry or productive, is presented separately from other respiratory symptoms due to its potential relation to quitting smoking.
Sleep disturbance (Psychiatric disorders) | 5 (5) | 6 (6) | 4 (4) | 3 (3) — Mild sleep disturbance (difficulty falling asleep, vivid dreams, waking in the night).
Gastrointestinal symptoms (Gastrointestinal disorders) | 5 (6) | 1 (1) | 1 (1) | 1 (1) — Heartburn, nausea, abdominal pain or cramping.
Headache (General disorders) | 4 (5) | 3 (3) | 1 (1) | 2 (3) — Headaches, including migraine headaches.
Skin irritation, rash, or pain (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 1 (1) | 4 (4) — Transdermal nicotine patches were provided to all participants and skin irritation, redness, rash, or discomfort at the patch site was reported by some participants.
Dizziness or lightheadedness (General disorders) | 4 (4) | 2 (2) | 0 (0) | 2 (2) — Feeling dizzy, lightheaded, or faint.
Fatigue (General disorders) | 3 (3) | 2 (3) | 0 (0) | 0 (0) — Tiredness, fatigue, sleepiness.

LIMITATIONS AND CAVEATS:
The sample comprised adult treatment-seeking smokers who met inclusion criteria and were willing to participate in a randomized controlled trial involving intensive assessment and offering substantial compensation.

The degree to which results will generalize to medically or mentally ill smokers is unknown.

Neither participants nor researchers were blind to condition assignment. All abstinence outcomes were based on self-report rather than biochemical verification.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Informed Consent Form (2013-01-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT01368653/ICF_000.pdf